CLINICAL TRIAL: NCT01698008
Title: Effect of Mobile Phone Telemedicine on Diabetes Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0396-12-FB
Record Dates: First submitted 2012-09-28; First posted 2012-10-02 (Estimated); Results first posted 2018-11-02 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: One group is standard of care. The other is given the opportunity to use a new mobile app for reporting blood sugars.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile application Diabetes Doctor (Experimental): The intervention group will send in blood glucoses once a month using the mobile phone app, Diabetes Doctor. All subjects will be evaluated at initial, 3 month, and 6 month visits. They will receive HbA1c on each visit. After 3 months, a Diabetes Quality of Life (QOL) survey will be completed. A Usability and Satisfaction of Diabetes Doctor (USDD) survey will also be obtained. At the 3 month visit, they will also be given the chance to discontinue the mobile app and switch to standard of care. At 6 months, all mobile app users will complete the USDD and satisfaction and QOL survey. If they are not using the mobile app, then they will complete the QOL survey.
  Interventions: Other: Diabetes Doctor Mobile app
- Standard of Care (No Intervention): The standard of care arm will not use the mobile application Diabetes Doctor to communicate with their physician about their blood sugars. They will attend clinic visits and have evaluations initially, and at 3 and 6 months. They will also receive a HbAIc at each visit. They will do the same QOL survey at 3 months. At 6 months, they will be given the QOL survey.

INTERVENTIONS:
Other: Diabetes Doctor Mobile app — Diabetes Doctor is a mobile application software. The mobile phone application allows a subject to register blood glucose values obtained from their fingerstick glucose meter readings, the type and amount of insulin they are administering, any notes they would like to document, and the date and time of each entry. All data will be entered by the subject manually. The data will be submitted through encryption coded private servers and can be retrievable by a physician on a password protected website for privacy. A physician will evaluate this information to recommend a change of the subject's insulin regimen. The recommended insulin regimen will be delivered to the patient using the same website and received by the subject on the same mobile application software.
  Arms: Mobile application Diabetes Doctor

SUMMARY:
Adult patients with diabetes on insulin are eligible for the study. They will be randomized to a group using standard of care communication and a group using an I phone intervention.

DETAILED DESCRIPTION:
Type 1 or type 2 diabetes mellitus subjects who know how to operate and own an iPhone, are between the age of 19 to 75, and are on a basal/bolus insulin regimen will be included in the study. Subjects will be randomized to two groups - iPhone versus standard of care and seen in our clinic at an initial/baseline and three month clinical visit. The control group will e-mail, fax, or call their blood glucose log results once a month for an insulin regimen adjustment through verbal communication with a certified diabetic educator once a month as is already implemented at the Diabetes Center. This group will be compared to the intervention group who will submit their blood glucose log results through an iPhone mobile application, called Diabetes Doctor, once a month for an insulin regimen adjustment by a physician with a text message response. The two groups will have their HbA1c, hypoglycemic events, blood glucose dispersion compliance, quality of life, usability and satisfaction with the use of a mobile application will be assessed at each visit with surveys.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or type 2 Diabetes Mellitus on insulin basal/bolus injection
* Own and are able to operate an iPhone

Exclusion Criteria:

* Type 2 diabetics using only oral medications
* Do not own or know how to operate an iPhone

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-01-28 (Actual); Primary Completion 2013-09-25 (Actual); Study Completion 2013-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Whitney S Goldner, MD, Principal Investigator — University of Nebraska
Locations (1):
- The University of Nebraska Medical Center, Omaha, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Mobile Application Diabetes Doctor: This group was given the opportunity to use the mobile app: Diabetes Doctor to send in blood sugars to communicate with their physician.
- Standard of Care Group: This group continued to communicate with their physician regarding their blood sugars as per standard of care and routine clinic follow ups. No intervention was made.
Period: Overall Study
Arm/Group | Mobile Application Diabetes Doctor | Standard of Care Group
Started | 3 | 2
Completed | 2 | 0
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Population: All patients have type 1 diabetes.
Groups:
- Mobile Application Diabetes Doctor: The intervention group sent blood glucoses once a month using the mobile phone app, Diabetes Doctor. Subjects were seen at initial, 3 month, and 6 month visits. They received HbA1c on each visit. After 3 months, a Diabetes Quality of Life (QOL)survey was completed. A Usability and Satisfaction of Diabetes Doctor (USDD) survey was given to assess use of the mobile app. At the 3 month interval the control group will be given the opportunity to use the mobile application. QOL and USDD was given at the conclusion of the study.
- Standard of Care Group: This group did not use the mobile app to communicate with their physician about their blood sugars. They continued with their current care.
- Total: Total of all reporting groups
Arm/Group | Mobile Application Diabetes Doctor | Standard of Care Group | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Evidence for Improved Diabetic Care With Mobile Phone Application Use
Description: Satisfaction and usability was evaluated with a survey for those subjects who used the mobile phone application at the 3 and 6 months period.
Time Frame: Six months
Population: Participants withdrew from study in standard of care group
Measure: Count of Participants; unit: Participants
Groups:
- Mobile Application Diabetes Doctor: This group was given the opportunity to use the mobile app Diabetes Doctor to communicate with their physician about their blood sugars.
- Standard of Care: This group followed standard of care, did not use the mobile app Diabetes Doctor.
Arm/Group | Mobile Application Diabetes Doctor | Standard of Care
Number analyzed (Participants) | 2 | 0
Participants | 2 | 0

ADVERSE EVENTS:
Time Frame: The data were collected for the duration of the study, 6 months.
Groups:
- Mobile Application Diabetes Doctor: This group used the mobile app Diabetes Doctor to communicate with their physicians about their blood sugars.
- Standard of Care: This group did not use the mobile app Diabetes Doctor to communicate with their physicians.
Arm/Group | Mobile Application Diabetes Doctor | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 0/3 | 0/2

LIMITATIONS AND CAVEATS:
Overall, there were difficulties with this study. We only had a small number of patients interested in participating and those that were given standard of care treatment did not continue on with the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes